CLINICAL TRIAL: NCT00265096
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Trial of Golimumab, a Fully Human Anti-TNFa MonoclonalAntibody, Administered Subcutaneously in Subjects With Active Psoriatic Arthritis
Brief Title: A Study of the Safety and Efficacy of Golimumab in Patients With Active Psoriatic Arthritis
Acronym: GO-REVEAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR006340; C0524T08 (Other: Centocor)
Record Dates: First submitted 2005-12-12; First posted 2005-12-14 (Estimated); Results first posted 2012-04-16 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Arthritis, Psoriatic
Keywords: Psoriatic Arthritis; Spondyloarthritis; Spondyloarthropathy; subcutaneous injection
MeSH Terms: conditions — Arthritis, Psoriatic; Spondylarthritis; Spondylarthropathies | interventions — golimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 002 (Experimental): golimumab 50 mg sc injs every 4 wks from wk 0 thru 5 yrs (unless early escape at wk 16); golimumab - if early escape, 100mg sc injection every 4 wks beginning wk 16 up to 5 yrs; golimumab - Dr's discretion after unblinding, dose adjust from 50 to 100mg
  Interventions: Biological: golimumab
- 001 (Experimental): Placebo; golimumab SC injections ever 4 wks thru Wk 20 (unless early escape at wk 16); golimumab - if early escape, 50mg sc injection from wk 16 up to 5 yrs; golimumab -50mg sc injection beginning Wk 24 up to 5 yrs (unless early escape); golimumab - Dr's discretion after unblinding, dose adjust from 50 to 100 mg
  Interventions: Biological: Placebo; golimumab
- 003 (Experimental): golimumab 100 mg sc injections every 4 wks from wk 0 up to 5 yrs
  Interventions: Biological: golimumab

INTERVENTIONS:
Biological: golimumab — 50 mg sc injs every 4 wks from wk 0 thru 5 yrs (unless early escape at wk 16); golimumab - if early escape, 100mg sc injection every 4 wks beginning wk 16 up to 5 yrs; golimumab - Dr's discretion after unblinding, dose adjust from 50 to 100mg
  Arms: 002
Biological: Placebo; golimumab — SC injections ever 4 wks thru Wk 20 (unless early escape at wk 16); golimumab - if early escape, 50mg sc injection from wk 16 up to 5 yrs; golimumab -50mg sc injection beginning Wk 24 up to 5 yrs (unless early escape); golimumab - Dr's discretion after unblinding, dose adjust from 50 to 100 mg
  Arms: 001
Biological: golimumab — 100 mg sc injections every 4 wks from wk 0 up to 5 yrs
  Arms: 003

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy (improvement of signs and symptoms) of subcutaneous (under the skin) injections of golimumab for the treatment of active psoriatic arthritis (PsA). Efficacy will be measured by reduction in the signs and symptoms of active PsA, including effects on joint pain and swelling, changes on x-ray related to joint damage, psoriasis skin lesions, physical function, and quality of life.

DETAILED DESCRIPTION:
Anti-tumor necrosis factor (TNF) agents have been shown to be effective in improving arthritis and psoriasis symptoms in patients with active psoriatic arthritis. Golimumab is a new anti-TNFa agent. This is a multicenter, randomized (patients are assigned different treatments based on chance), double-blind (neither the patient nor the physician knows whether drug or placebo is being taken, or at what dosage), placebo-controlled, parallel group study comparing safety and efficacy of golimumab 50mg, golimumab 100mg, and placebo subcutaneous injections administered every 4 weeks, in subjects with active PsA. The total duration of treatment is approximately 5 years. In the first portion of the study, some patients will be randomly assigned to receive placebo treatment through the Week 20 injection; others will be assigned to golimumab 50mg or golimumab 100mg groups through the Week 20 injection. There is an "early escape" at Week 16 in the study whereby patients who meet criteria for minimal improvement in their joints will be switched to golimumab if they were on placebo, or have the golimumab dose increased if they were originally assigned to the golimumab 50mg group. At Week 24, the placebo group subjects will switch to golimumab 50mg injections, and all patients will continue receiving in a blinded manner either 50 or 100mg golimumab injections every 4 weeks until the first 52 weeks of data are fully collected on all the subjects (database lock). After this 52-week database lock, everyone will be unblinded to the golimumab dose, and continue to receive golimumab treatment through Week 252 as part of a long-term extension phase of the study, with options for adjusting concomitant PsA medications and/or increasing the dose of golimumab. The study hypothesis is that golimumab will be more effective than placebo both in terms of reducing the signs and symptoms of PsA, as measured by the American College of Rheumatology (ACR) 20 response at Week 14, and inhibiting the amount of damage due to PsA seen on x-rays of the hand and feet at Week 24, while maintaining an acceptable safety profile. Golimumab 50mg, Golimumab 100mg, or placebo injected under the skin every 4 weeks at Weeks 0, 4, 8, 12, 16, and 20, followed by injections of either Golimumab 50mg or Golimumab 100mg every 4 weeks, for approximately 5 years total duration from the time of the first study agent injection.

ELIGIBILITY:
Inclusion Criteria:

* Psoriatic arthritis (PsA) diagnosed > 6months prior
* Active PsA at the time of screening and at baseline visits, with >= 3 swollen joints and >= 3 tender joints
* Have at least 1 of the PsA subsets (DIP joint arthritis, polyarticular arthritis without rheumatoid nodules, arthritis mutilans, asymmetric peripheral arthritis, or spondylitis with peripheral arthritis)
* Active plaque psoriasis with a lesion >= 2cm in diameter
* Active arthritis despite current disease modifying anti-rheumatic drug (DMARD) or nonsteroidal anti-inflammatory drug (NSAID) therapy
* Stable doses of methotrexate, low-dose corticosteroids, and NSAIDs are permitted.

Exclusion Criteria:

* No prior treatment with biologic anti-TNF agents (infliximab, etanercept, adalimumab)
* No treatment with alefacept or efalizumab within 3 months prior to the first study drug injection
* No DMARDs other than methotrexate, or immunosuppressive drugs within 4 weeks prior to the first study drug injection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2005-12; Primary Completion 2007-05 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.
Locations (51):
- United States (18):
  - Huntsville, Alabama
  - La Jolla, California
  - Upland, California
  - Aventura, Florida
  - Coeur d'Alene, Idaho
  - Kansas City, Kansas
  - Wheaton, Maryland
  - Worcester, Massachusetts
  - Omaha, Nebraska
  - Cincinnati, Ohio
  - Mayfield, Ohio
  - Lake Oswego, Oregon
  - Portland, Oregon
  - Duncansville, Pennsylvania
  - West Reading, Pennsylvania
  - Houston, Texas
  - Edmonds, Washington
  - Seattle, Washington
- Belgium (5):
  - Brussels
  - Ghent
  - Leuven
  - Liège
  - Merksem
- Canada (15):
  - Victoria, British Columbia
  - Winnipeg, Manitoba
  - St. John's, Newfoundland and Labrador
  - North Bay, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Waterloo, Ontario
  - Montreal, Quebec
  - Sainte-Foy, Quebec
  - Sante Foy, Quebec
  - Claire
  - Hamilton Ontario
  - Newmarket
  - Saskatoon
  - Vancouver
- Poland (7):
  - Bialystok
  - Elblag
  - Kalisz
  - Poznan
  - Szczecin
  - Torun
  - Warsaw
- Spain (2):
  - Santiago de Compostela
  - Valencia
- United Kingdom (4):
  - Glasgow
  - London
  - Middlesbrough
  - Wigan

REFERENCES:
- [Derived] Leu JH, Adedokun OJ, Gargano C, Hsia EC, Xu Z, Shankar G. Immunogenicity of golimumab and its clinical relevance in patients with rheumatoid arthritis, psoriatic arthritis and ankylosing spondylitis. Rheumatology (Oxford). 2019 Mar 1;58(3):441-446. doi: 10.1093/rheumatology/key309. PMID 30412238
- [Derived] Kay J, Fleischmann R, Keystone E, Hsia EC, Hsu B, Zhou Y, Goldstein N, Braun J. Five-year Safety Data from 5 Clinical Trials of Subcutaneous Golimumab in Patients with Rheumatoid Arthritis, Psoriatic Arthritis, and Ankylosing Spondylitis. J Rheumatol. 2016 Dec;43(12):2120-2130. doi: 10.3899/jrheum.160420. Epub 2016 Nov 1. PMID 27803138
- [Derived] Aletaha D, Alasti F, Smolen JS. Disease activity states of the DAPSA, a psoriatic arthritis specific instrument, are valid against functional status and structural progression. Ann Rheum Dis. 2017 Feb;76(2):418-421. doi: 10.1136/annrheumdis-2016-209511. Epub 2016 Jul 25. PMID 27457512
- [Derived] Kavanaugh A, van der Heijde D, Beutler A, Gladman D, Mease P, Krueger GG, McInnes IB, Helliwell P, Coates LC, Xu S. Radiographic Progression of Patients With Psoriatic Arthritis Who Achieve Minimal Disease Activity in Response to Golimumab Therapy: Results Through 5 Years of a Randomized, Placebo-Controlled Study. Arthritis Care Res (Hoboken). 2016 Feb;68(2):267-74. doi: 10.1002/acr.22576. PMID 25779603
- [Derived] Kavanaugh A, McInnes IB, Mease P, Krueger GG, Gladman D, van der Heijde D, Zhou Y, Lu J, Leu JH, Goldstein N, Beutler A. Clinical efficacy, radiographic and safety findings through 5 years of subcutaneous golimumab treatment in patients with active psoriatic arthritis: results from a long-term extension of a randomised, placebo-controlled trial (the GO-REVEAL study). Ann Rheum Dis. 2014 Sep;73(9):1689-94. doi: 10.1136/annrheumdis-2013-204902. Epub 2014 Apr 19. PMID 24748630
- [Derived] Helliwell PS, Kavanaugh A. Comparison of composite measures of disease activity in psoriatic arthritis using data from an interventional study with golimumab. Arthritis Care Res (Hoboken). 2014 May;66(5):749-56. doi: 10.1002/acr.22204. PMID 24127416
- [Derived] Kavanaugh A, McInnes IB, Krueger GG, Gladman D, Beutler A, Gathany T, Mack M, Tandon N, Han C, Mease P. Patient-reported outcomes and the association with clinical response in patients with active psoriatic arthritis treated with golimumab: findings through 2 years of a phase III, multicenter, randomized, double-blind, placebo-controlled trial. Arthritis Care Res (Hoboken). 2013 Oct;65(10):1666-73. doi: 10.1002/acr.22044. PMID 23666608
- [Derived] Kavanaugh A, van der Heijde D, McInnes IB, Mease P, Krueger GG, Gladman DD, Gomez-Reino J, Papp K, Baratelle A, Xu W, Mudivarthy S, Mack M, Rahman MU, Xu Z, Zrubek J, Beutler A. Golimumab in psoriatic arthritis: one-year clinical efficacy, radiographic, and safety results from a phase III, randomized, placebo-controlled trial. Arthritis Rheum. 2012 Aug;64(8):2504-17. doi: 10.1002/art.34436. PMID 22378566

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 405 patients were randomized at 57 centers: 35 in North America (17 in the United States and 18 in Canada) and 22 in Europe (5 in Belgium, 10 in Poland, 3 in Spain, and 4 in the United Kingdom). The first patient was enrolled on 12 Dec 2005. The date of the last patient visit for the week (Wk) 24 reporting period was 14 May 2007.
Groups:
- Group 1: Placebo: Group 1: Placebo Placebo subcutaneous (SC) injections every 4 weeks from week (Wk) 0 through Wk 20 (unless early escape at Wk 16); golimumab - if early escape, 50 mg SC injection from Wk 16 up to 5 years (yrs); golimumab - 50 mg SC injection beginning Wk 24 up to 5 yrs (unless early escape); golimumab - Doctor's (Dr's) discretion after unblinding (last patient completes the Wk 52 evaluation and database is locked), dose adjust from 50 to 100 mg.
- Group 2: Golimumab 50 mg: Golimumab 50 mg SC injections every 4 weeks from Wk 0 through 5 yrs (unless early escape at Wk 16); golimumab - if early escape, 100 mg SC injection every 4 weeks beginning Wk 16 up to 5 yrs; golimumab - Dr's discretion after unblinding (last patient completes the Wk 52 evaluation and database is locked), dose adjust from 50 to 100 mg.
- Group 3: Golimumab 100 mg: Golimumab 100 mg SC injections every 4 weeks from Wk 0 up to 5 yrs.
Period: Overall Study
Arm/Group | Group 1: Placebo | Group 2: Golimumab 50 mg | Group 3: Golimumab 100 mg
Started | 113 | 146 | 146
Completed | 77 (Indicates number of patients that were continuing SC study agent at Wk 24) | 95 (Indicates number of patients that were continuing SC study agent at Wk 24) | 107 (Indicates number of patients that were continuing SC study agent at Wk 24)
Not Completed | 36 | 51 | 39
Not completed — Adverse Event | 14 | 18 | 18
Not completed — Lost to Follow-up | 2 | 5 | 3
Not completed — Death | 0 | 1 | 2
Not completed — Unsatisfactory therapeutic effect | 9 | 8 | 6
Not completed — Other | 11 | 19 | 10

BASELINE CHARACTERISTICS:
Groups:
- Group 1: Placebo: Placebo subcutaneous (SC) injections every 4 weeks from week (Wk) 0 through Wk 20 (unless early escape at Wk 16); golimumab - if early escape, 50 mg SC injection from Wk 16 up to 5 years (yrs); golimumab - 50 mg SC injection beginning Wk 24 up to 5 yrs (unless early escape); golimumab - Doctor's (Dr's) discretion after unblinding (last patient completes the Wk 52 evaluation and database is locked), dose adjust from 50 to 100 mg.
- Total: Total of all reporting groups
Arm/Group | Group 1: Placebo | Group 2: Golimumab 50 mg | Group 3: Golimumab 100 mg | Total
Number analyzed (Participants) | 113 | 146 | 146 | 405
Age Continuous [Mean (Standard Deviation); unit: years] | 47 (10.56) | 45.7 (10.7) | 48.2 (10.93) | 47 (10.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 57 | 60 | 161
  Male | 69 | 89 | 86 | 244

OUTCOME MEASURES:

1. Primary Outcome: American College of Rheumatology (ACR) 20 Response at Week 14
Description: ACR 20 response is an improvement of >= 20% from baseline (baseline measurement is defined as the closest measurement taken prior to or at the time of the initiation of study medication administration) in both the tender and swollen joint count and in at least 3 of the 5 assessments (Patient's assessment of pain, Patient's global assessment of disease activity, Physician's global assessment of disease activity Visual Analogue Scale [VAS], Health Assessment Questionnaire [HAQ] and C-reactive protein [CRP])
Time Frame: Baseline (Week 0), Week 4, Week 8 and Week 14
Population: Intention to treat (ITT). Patients considered non-responder if used any pre-specified prohibited medications or discontinued subcutaneous (SC) study agent due to lack of efficacy. Missing ACR components at Week 14 were imputed by Last Observation Carried Forward (LOCF) unless all ACR components are missing in which case considered non-responders.
Measure: Number; unit: Participants
Groups:
- Group I: Placebo: Placebo subcutaneous (SC) injections every 4 weeks from week (Wk) 0 through Wk 20 (unless early escape at Wk 16); golimumab - if early escape, 50 mg SC injection from Wk 16 up to 5 years (yrs); golimumab - 50 mg SC injection beginning Wk 24 up to 5 yrs (unless early escape); golimumab - Doctor's (Dr's) discretion after unblinding (last patient completes the Wk 52 evaluation and database is locked), dose adjust from 50 to 100 mg.
- Group II: Golimumab 50 mg: Golimumab 50 mg SC injections every 4 weeks from Wk 0 through 5 yrs (unless early escape at Wk 16); golimumab - if early escape, 100 mg SC injection every 4 weeks beginning Wk 16 up to 5 yrs; golimumab - Dr's discretion after unblinding (last patient completes the Wk 52 evaluation and database is locked), dose adjust from 50 to 100 mg.
- Group III: Golimumab 100 mg: Golimumab 100 mg SC injections every 4 weeks from Wk 0 up to 5 yrs.
- Combined: Group II & III: Combines Group II (golimumab 50 mg) and Group III (golimumab 100 mg).
Arm/Group | Group I: Placebo | Group II: Golimumab 50 mg | Group III: Golimumab 100 mg | Combined: Group II & III
Number analyzed (Participants) | 113 | 146 | 146 | 292
Participants | 10 | 74 | 66 | 140
Statistical Analysis 1: Comparison: Group I: Placebo vs Combined: Group II & III; Null Hypothesis: No difference in ACR 20 response comparing Groups I vs II and Groups I vs III. Sample size (n=396; 110 placebo, 286 combined golimumab) provided >98% power to detect a significant difference (alpha=0.05) in ACR 20 response between treatment groups, assuming equal proportions of subjects receiving methotrexate (MTX) at baseline and the difference in ACR 20 response of 27% in subjects without MTX and 17-27% in subjects with MTX, between placebo and combined golimumab groups; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — The positive test is concluded if there is a significant difference between combined golimumab and placebo groups and at least one of the pair-wise conparisons at 0.05 level; Cochran-Mantel-Haenszel (CMH) with stratification (stratified by baseline MTX usage)
Statistical Analysis 2: Comparison: Group I: Placebo vs Group II: Golimumab 50 mg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) with stratification (stratified by baseline MTX usage)
Statistical Analysis 3: Comparison: Group I: Placebo vs Group III: Golimumab 100 mg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) with stratification (stratified by baseline MTX usage)

2. Secondary Outcome: Psoriasis Area and Severity Index (PASI) 75 Response at Week 14 in a Subset of Patients With ≥ 3 Percent Body Surface Area (BSA) Psoriasis Skin Involvement at Baseline
Description: Number of patients (randomized patients with >= 3 percent Body Surface Area [BSA] psoriasis skin involvement at baseline) with Psoriasis Area and Severity Index (PASI) 75 response at Week 14. PASI is the widely used tool for the measurement of severity of psoriasis. PASI combines the assessment of the severity of lesions and the area affected into a single score in the range of 0 to 72. Zero (0) means no disease and 72 means maximal disease. PASI 75 Response at Week 14 means reduction in PASI score by 75 percent at Week 14.
Time Frame: Baseline, Week 4, Week 8 and Week 14
Population: In a subset of patients with ≥ 3 percent body surface area (BSA) psoriasis skin involvement at baseline. Missing scores were imputed by Last Observation Carried Forward (LOCF).
Measure: Number; unit: Participants
Groups:
- Group III: Golimumab 100 mg: Golimumab 100 mg SC injections every 4 wks from Wk 0 up to 5 yrs.
Arm/Group | Group I: Placebo | Group II: Golimumab 50 mg | Group III: Golimumab 100 mg | Combined: Group II & III
Number analyzed (Participants) | 79 | 109 | 108 | 217
Participants | 2 | 44 | 63 | 107
Statistical Analysis 1: Comparison: Group I: Placebo vs Combined: Group II & III; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) with stratification (stratified by baseline MTX usage)
Statistical Analysis 2: Comparison: Group I: Placebo vs Group II: Golimumab 50 mg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) with stratification (stratified by baseline MTX usage)
Statistical Analysis 3: Comparison: Group I: Placebo vs Group III: Golimumab 100 mg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) with stratification (stratified by baseline MTX usage)

3. Secondary Outcome: Improvement From Baseline in Health Assessment Questionnaire Scores at Week 24
Description: Summary of improvement from baseline in Health Assessment Questionnaire (HAQ) score at Week (Wk) 24. This 20-question instrument assesses the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living). Responses in each functional area are scored from 0, indicating no difficulty, to 3, indicating inability to perform a task in that area based on the worst score from the questions that pertain to that task. The HAQ score is determined by the average of the 8 scores.
Time Frame: Baseline, Week 4, Week 8, Week 14, Week 16, Week 20 and Week 24
Population: Intention to treat (ITT). Missing scores were imputed by LOCF. Week (Wk) 16 scores were used for patients with change in study treatment. Week 16 HAQ scores were used for patients with change in study treatment.
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | Group I: Placebo | Group II: Golimumab 50 mg | Group III: Golimumab 100 mg | Combined: Group II & III
Number analyzed (Participants) | 113 | 146 | 146 | 292
scores on a scale | 0.0000 (0.48796) [-0.2500 to 0.2500] | 0.2500 (0.55215) [0.0000 to 0.6250] | 0.3750 (0.50329) [0.0000 to 0.6250] | 0.2500 (0.52811) [0.0000 to 0.6250]
Statistical Analysis 1: Comparison: Group I: Placebo vs Combined: Group II & III; Test type: Superiority or Other; p < 0.001, ANOVA on van der Waerden normal scores; With 2 factors (treatment group and subject's baseline Methotrexate (MTX) usage)
Statistical Analysis 2: Comparison: Group I: Placebo vs Group II: Golimumab 50 mg; Test type: Superiority or Other; p < 0.001, ANOVA on van der Waerden normal scores; With 2 factors (treatment group and subject's baseline MTX usage)
Statistical Analysis 3: Comparison: Group I: Placebo vs Group III: Golimumab 100 mg; Test type: Superiority or Other; p < 0.001, ANOVA on van der Waerden normal scores; With 2 factors (treatment group and subject's baseline MTX usage)

4. Secondary Outcome: Change From Baseline in the Physical Component Summary Score of the 36-item Short Form Health Survey at Week 14
Description: The short form health survey (SF-36) is a well-validated and widely used quality-of-life instrument employed in numerous disease states. It is a self-administered survey that measures eight domains of health including: physical functioning, role limitations due to physical health (role-physical), bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems (role-emotional) and general mental health. Scoring of the SF-36 was based on the SF-36 Manual and Interpretation Guide. Worst value is 0 and best value is 100.
Time Frame: Baseline and Week 14
Population: Intention to treat (ITT). Missing scores were imputed by Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Group I: Placebo | Group II: Golimumab 50 mg | Group III: Golimumab 100 mg | Combined: Group II & III
Number analyzed (Participants) | 113 | 146 | 146 | 292
scores on a scale | 0.63 (7.676) | 6.53 (8.882) | 7.85 (9.547) | 7.19 (9.229)
Statistical Analysis 1: Comparison: Group I: Placebo vs Combined: Group II & III; Test type: Superiority or Other; p < 0.001, ANOVA on van der Waerden normal scores; With 2 factors (treatment and subject's baseline Methotrexate (MTX) usage)
Statistical Analysis 2: Comparison: Group I: Placebo vs Group II: Golimumab 50 mg; Test type: Superiority or Other; p < 0.001, ANOVA on van der Waerden normal scores; With 2 factors (with treatment and subject's baseline MTX usage)
Statistical Analysis 3: Comparison: Group I: Placebo vs Group III: Golimumab 100 mg; Test type: Superiority or Other; p < 0.001, ANOVA on van der Waerden normal scores; With 2 factors (treatment and subject's baseline MTX usage)

5. Primary Outcome: Change From Baseline in Total Radiographic Scores of the Hands and Feet at Week 24
Description: Summary of change from baseline in total van der Heijde-Sharp (vdH-S) score of the hands and feet, as modified for psoriatic arthritis, at Week 24. The vdH-S score is the sum of joint erosion score and joint-space narrowing (JSN) score. The total score ranges from 0 to 528 with higher scores indicating more joint damage. For the change from baseline, positive values show an increase in damage.
Time Frame: Baseline and Week 24
Population: Intent-to-treat analysis.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Group I: Placebo | Group II: Golimumab 50 mg | Group III: Golimumab 100 mg | Combined: Group II & III
Number analyzed (Participants) | 113 | 146 | 146 | 292
Scores on a scale | 0.27 (1.259) | -0.16 (1.309) | -0.02 (1.322) | -0.09 (1.315)
Statistical Analysis 1: Comparison: Group I: Placebo vs Combined: Group II & III; Null Hypothesis: There is no difference in change from baseline among 3 treatment groups. Sample size (n=396, 110 placebo, 286 combined golimumab) provided >93% power to detect a significant difference (alpha=0.05) in change from baseline between treatment groups, assuming 50% of subjects received MTX at baseline, and mean change from baseline for combined golimumab of 0, and a mean increase for placebo of 0.1 in subjects who received MTX at baseline and 0.6 in subjects who did not receive MTX; Test type: Superiority or Other; p = 0.015, ANOVA — The test was not to be performed if the test of ACR 20 at Week 24 was not significant; Analysis of Variance (ANOVA) on van der Waerden scores with 2 factors: treatment group and participant's baseline methotrexate (MTX) usage
Statistical Analysis 2: Comparison: Group I: Placebo vs Group II: Golimumab 50 mg; Test type: Superiority or Other; p = 0.011, ANOVA — The test was not to be performed if the test of ACR 20 at Week 24 was not significant; ANOVA on van der Waerden scores with 2 factors: treatment group and participant's baseline Methotrexate (MTX) usage
Statistical Analysis 3: Comparison: Group I: Placebo vs Group III: Golimumab 100 mg; Test type: Superiority or Other; p = 0.086, ANOVA — The test was not to be performed if the test of ACR 20 at Week 24 was not significant; ANOVA on van der Waerden scores with 2 factors: treatment group and participant's baseline Methotrexate (MTX) usage

6. Secondary Outcome: American College of Rheumatology 20 at Week 24
Description: Number of Patients who achieved an American College of Rheumatology (ACR) 20 response at Week (Wk) 24.
  ACR 20 response is an improvement of >= 20% from baseline in both the tender and swollen joint count and in at least 3 of the 5 assessments (Patient's assessment of pain, Patient's global assessment of disease activity, Physician's global assessment of disease activity Visual Analogue Scale [VAS], Health Assessment Questionnaire [HAQ] and C-reactive protein [CRP])
Time Frame: Baseline, Week 4, Week 8, Week 14, Week 16, Week 20 and Week 24
Population: ITT. Patients considered non-responder if used any pre-specified prohibited medications or discontinued SC study agent due to lack of efficacy. Missing ACR components were imputed by LOCF unless all ACR components are missing in which case considered non-responders. Wk 16 ACR response was used for patients with change in study treatment.
Measure: Number; unit: P a r t i c ip an t s
Arm/Group | Group I: Placebo | Group II: Golimumab 50 mg | Group III: Golimumab 100 mg | Combined: Group II & III
Number analyzed (Participants) | 113 | 146 | 146 | 292
P a r t i c ip an t s | 14 | 76 | 89 | 165
Statistical Analysis 1: Comparison: Group I: Placebo vs Combined: Group II & III; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) with stratification (stratified by baseline Methotrexate (MTX) usage)
Statistical Analysis 2: Comparison: Group I: Placebo vs Group II: Golimumab 50 mg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) with stratification (stratified by baseline MTX usage)
Statistical Analysis 3: Comparison: Group I: Placebo vs Group III: Golimumab 100 mg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) with stratification (stratified by baseline MTX usage)

ADVERSE EVENTS:
Description: The number of participants reported at risk for adverse events (AEs) in each treatment (tx) group is based on actual tx received during the study and may differ from the number of participants who started tx in the study. Participants may be counted more than once in the analysis of AEs if they received tx at more than one dose level in the study.
Groups:
- Group 1: Golimumab 50 mg: Subjects who were treated with Golimumab and received Golimumab 50 mg injections only.
- Group 2: Golimumab 100 mg: Subjects who were treated with Golimumab and received Golimumab 100 mg injections only.
- Group 3: Golimumab 50 and 100 mg: Subjects who were treated with Golimumab and received at least one injection of both Golimumab 50 mg and Golimumab 100 mg.
Arm/Group | Group 1: Golimumab 50 mg | Group 2: Golimumab 100 mg | Group 3: Golimumab 50 and 100 mg
Serious Adverse Events (participants affected / at risk) | 29/139 | 25/109 | 29/146
Other Adverse Events (participants affected / at risk) | 107/139 | 91/109 | 113/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Golimumab 50 mg (N=139) | Group 2: Golimumab 100 mg (N=109) | Group 3: Golimumab 50 and 100 mg (N=146)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Acute Left Ventricular Failure (Cardiac disorders) | 0 | 0 | 1
Acute Myocardial Infarction (Cardiac disorders) | 0 | 1 | 0
Cardiac Failure Congestive (Cardiac disorders) | 0 | 1 | 0
Coronary Artery Disease (Cardiac disorders) | 1 | 0 | 0
Coronary Artery Occlusion (Cardiac disorders) | 0 | 0 | 1
Myocardial Infarction (Cardiac disorders) | 4 | 0 | 1
Myocardial Ischaemia (Cardiac disorders) | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1
Erosive Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1
Irritable Bowel Syndrome (Gastrointestinal disorders) | 0 | 0 | 1
Oesophageal Pain (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Accidental Death (General disorders) | 1 | 1 | 0
Chest Pain (General disorders) | 0 | 0 | 2
Death (General disorders) | 0 | 1 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 2 | 0
Abscess (Infections and infestations) | 2 | 0 | 0
Arthritis Bacterial (Infections and infestations) | 0 | 0 | 1
Bartholin's Abscess (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 1
Eye Infection Toxoplasmal (Infections and infestations) | 0 | 1 | 0
Histoplasmosis (Infections and infestations) | 0 | 1 | 0
Lung Abscess (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 2
Pneumonia Legionella (Infections and infestations) | 0 | 0 | 1
Pyelonephritis Acute (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Streptococcal Sepsis (Infections and infestations) | 0 | 0 | 1
Tuberculosis (Infections and infestations) | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Delayed Recovery from Anaesthesia (Injury, poisoning and procedural complications) | 0 | 0 | 1
Limb Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tendon Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tibia Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Alanine Aminotransferase Increased (Investigations) | 1 | 0 | 0
Hepatic Enzyme Increased (Investigations) | 0 | 1 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Foot Deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Intervertebral Disc Disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Psoriatic Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4 | 3
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bladder Transitional Cell Carcinoma Stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Colon Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon Cancer Stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Oesophageal Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Renal Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Small Cell Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Small Cell Lung Cancer Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Squamous Cell Carcinoma of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 1 | 0
Balance Disorder (Nervous system disorders) | 0 | 1 | 0
Carotid Artery Stenosis (Nervous system disorders) | 0 | 0 | 1
Cervical Myelopathy (Nervous system disorders) | 0 | 0 | 1
Myelopathy (Nervous system disorders) | 1 | 0 | 0
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Alcoholism (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 1 | 0
Suicidal Ideation (Psychiatric disorders) | 0 | 0 | 1
Calculus Urinary (Renal and urinary disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Renal Colic (Renal and urinary disorders) | 1 | 0 | 0
Renal Failure (Renal and urinary disorders) | 1 | 0 | 0
Ovarian Cyst (Reproductive system and breast disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1
Thrombophlebitis Superficial (Vascular disorders) | 1 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Golimumab 50 mg (N=139) | Group 2: Golimumab 100 mg (N=109) | Group 3: Golimumab 50 and 100 mg (N=146)
Conjunctivitis (Eye disorders) | 8 | 3 | 2
Abdominal Pain (Gastrointestinal disorders) | 6 | 9 | 6
Diarrhoea (Gastrointestinal disorders) | 11 | 15 | 13
Dyspepsia (Gastrointestinal disorders) | 11 | 4 | 6
Nausea (Gastrointestinal disorders) | 6 | 7 | 9
Fatigue (General disorders) | 4 | 8 | 11
Injection Site Erythema (General disorders) | 12 | 13 | 7
Oedema Peripheral (General disorders) | 5 | 6 | 8
Bronchitis (Infections and infestations) | 18 | 11 | 18
Cellulitis (Infections and infestations) | 7 | 1 | 6
Ear Infection (Infections and infestations) | 2 | 8 | 8
Gastroenteritis (Infections and infestations) | 8 | 8 | 6
Influenza (Infections and infestations) | 10 | 7 | 8
Nasopharyngitis (Infections and infestations) | 23 | 28 | 31
Oral Herpes (Infections and infestations) | 9 | 5 | 4
Pharyngitis (Infections and infestations) | 7 | 5 | 13
Rhinitis (Infections and infestations) | 5 | 6 | 7
Sinusitis (Infections and infestations) | 18 | 13 | 20
Upper Respiratory Tract Infection (Infections and infestations) | 44 | 34 | 41
Urinary Tract Infection (Infections and infestations) | 10 | 12 | 6
Ligament Sprain (Injury, poisoning and procedural complications) | 3 | 5 | 11
Muscle Strain (Injury, poisoning and procedural complications) | 3 | 6 | 4
Alanine Aminotransferase Increased (Investigations) | 17 | 8 | 11
Aspartate Aminotransferase Increased (Investigations) | 11 | 5 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 | 10 | 14
Back Pain (Musculoskeletal and connective tissue disorders) | 18 | 18 | 22
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 | 6 | 2
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 6 | 7 | 6
Psoriatic Arthropathy (Musculoskeletal and connective tissue disorders) | 15 | 13 | 12
Tendonitis (Musculoskeletal and connective tissue disorders) | 11 | 3 | 5
Headache (Nervous system disorders) | 21 | 14 | 12
Sciatica (Nervous system disorders) | 2 | 6 | 4
Anxiety (Psychiatric disorders) | 7 | 2 | 2
Depression (Psychiatric disorders) | 8 | 7 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 8 | 12
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 7 | 8 | 6
Night Sweats (Skin and subcutaneous tissue disorders) | 8 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 0 | 3
Psoriasis (Skin and subcutaneous tissue disorders) | 11 | 6 | 15
Rash (Skin and subcutaneous tissue disorders) | 5 | 6 | 9
Hypertension (Vascular disorders) | 12 | 16 | 24

LIMITATIONS AND CAVEATS:
The count of patients with any nonserious adverse events (NAE) excludes patients who only had NAE that occurred in <=5% of patients. This information may vary from existing approved labeling and publications due to the requirement of this website.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, the only disclosure restriction on the PI is that the sponsor has 60 days to review results communications prior to public release and can embargo communications regarding trial results for a period that does not exceed 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.